CLINICAL TRIAL: NCT00739336
Title: Diabetes Prevention and Control in the Workplace: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: County of Onondaga, NYS (Unknown); NYS Department of Health (Unknown)
Responsible Party: Principal Investigator, Ruth Weinstock, Distinguished Service Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB#5657; NYSDOH Contract# C021750; Onondaga Cty,NY Contract#39407
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes mellitus; obesity; prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, 1 (Experimental): Intervention: Immediate 3 month program
  Interventions: Behavioral: Diabetes Prevention and Control
- A, 2 (No Intervention): Wait-List Control

INTERVENTIONS:
Behavioral: Diabetes Prevention and Control — The program will be delivered over 3 months in 12 one hour weekly mid-day sessions at the worksite. The curriculum has been adapted from the Diabetes Prevention Program, the National Diabetes Education Program and Conversation maps from Healthy Interactions Inc. Topics relate to healthy eating, physical activity, coping with disease and depression, and cardiovascular disease prevention. Additional topics may be included per feedback and need of the participants. After completion of the 3 month program, there will be monthly meetings.
  Arms: A, 1

SUMMARY:
This worksite program for Onondaga County employees is a pilot research study aimed at decreasing the risk of developing diabetes (or improving metabolic control for adults with diabetes). The main goal is to improve the nutrition and physical habits of the participants, and promote weight loss in those who are overweight. The investigators will also examine factors that predict participation in the program and influence a participant's outcome/success in the program.

ELIGIBILITY:
Inclusion Criteria:

* Adult employees of Onondaga County

Exclusion Criteria:

* Not an employee of Onondaga County
* Less than age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth S Weinstock, MD, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Barham K, West S, Trief P, Morrow C, Wade M, Weinstock RS. Diabetes prevention and control in the workplace: a pilot project for county employees. J Public Health Manag Pract. 2011 May-Jun;17(3):233-41. doi: 10.1097/PHH.0b013e3181fd4cf6. PMID 21464685

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: A 3 month program (12 one hour weekly sessions) that targets healthy diet, physical activity and stress reduction, and then a monthly maintenance program for up to 2 years.
- Control: This is a "wait control" group, This group will begin the program (described in A,1) after 3 months.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 21 | 24
Completed | 17 | 24
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: A 3 month program (12 one hour weekly sessions) that targets healthy diet, physical activity and stress reduction, and then a monthly maintenance program for up to 2 years.
  Diabetes Prevention and Control: The program will be delivered over 3 months in 12 one hour weekly mid-day sessions at the worksite. The curriculum has been adapted from the Diabetes Prevention Program, the National Diabetes Education Program and Conversation maps from Healthy Interactions Inc. Topics relate to healthy eating, physical activity, coping with disease and depression, and cardiovascular disease prevention. Additional topics may be included per feedback and need of the participants. After completion of the 3 month program, there will be monthly meetings.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (9.6) | 51.2 (6.4) | 51.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Weight loss in kg
Time Frame: 3 months
Population: Participants from the wait-list "Control" Arm have been combined in the "Intervention" Arm with those receiving the intervention immediately upon study entry for the purposes of this analysis.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 41 | 24
kg | -2.3 [-3.5 to -0.97] | 0.73 [0.17 to 1.28]
Statistical Analysis 1: Comparison: Intervention vs Control; Piecewise linear multilevel models with multiple observations nested within each participant were used. Random components (intercept, slope) were introduced into the model to account for dependence among measurements within a participant and assessed by nested model comparisons using the deviance statistic (difference in -2LL); Test type: Superiority or Other; p < 0.01, Mixed Models Analysis

2. Secondary Outcome: Fasting Glucose Level
Description: Fasting glucose (mg/dL)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 24
mg/dL | 107 (36) | 111 (36)

3. Secondary Outcome: Fasting Lipid Profile
Description: LDL-cholesterol (mg/dL)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 24
mg/dL | 126 (24) | 112 (34)

4. Secondary Outcome: Hemoglobin A1c
Description: hemoglobin A1c (%)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 24
percent | 6.2 (1.3) | 6.4 (1.3)

5. Secondary Outcome: Waist Circumference
Time Frame: baseline, 3, 6, 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Questionnaires
Time Frame: baseline, 3, 6, 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: Participants from the wait-list "Control" Arm have been combined in the "Intervention" Arm with those receiving the intervention immediately upon study entry for the purposes of Adverse Events collection.
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/24
Other Adverse Events (participants affected / at risk) | 0/45 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No